CLINICAL TRIAL: NCT01617018
Title: Systemic Treatment for Psoriasis Patients: A Prospective Multicentric Observational Cohort Study
Brief Title: Assessing the Long Term Effectiveness and Safety of Biotherapies in the Treatment of Cutaneous Psoriasis
Acronym: PSOBIOTEQ
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Health Products Safety Agency (Other Government); Société de Dermatologie Française (Other); Janssen, LP (Industry); Pfizer (Industry); AbbVie (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AOM09195; N° IRB00006477 (Other: EudraCTNumber)
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Psoriasis
Keywords: Psoriasis; Biological therapy; Methotrexate; Cyclosporine
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed group: Biotherapy
- Non-exposed group: Major conventional systemic therapy (methotrexate or cyclosporine)

SUMMARY:
PSOBIOTEQ is a national multicentric prospective cohort of cutaneous psoriasis patients receiving systemic treatment (biotherapy or DMARDs) for moderate to severe cutaneous psoriasis. It is resulting from the merging of two studies that share the same study population but address different objectives: PSOBIO, developed by academic dermatologists and epidemiologists and supported by the National Drug Agency (AGENCE NATIONALE DE SECURITE DU MEDICAMENT ET DES PRODUITS DE SANTE,ANSM) and the ministry of health (PHRC 2009) focusing on safety issues, and Pso-TEQ, developed by industrials at the request of the French Transparency Commission (HAUTE AUTORITE DE SANTE) focusing on utilisation issues.

The overall general objective of PSOBIO is to assess "in real life" the safety and efficacy of biotherapies in the treatment of cutaneous psoriasis in comparison with major conventional systemic therapy while Pso-TEQ has a descriptive objective concerning the modalities of use of biological therapies "in real life" and long-term benefit.

DETAILED DESCRIPTION:
PSOBIOTEQ is a national multicentric prospective cohort, including patients receiving systemic treatment (biotherapy or DMARDs) for moderate to severe cutaneous psoriasis.

The exposure of interest is the exposure to a biological therapy: infliximab, adalimumab, etanercept, ustekinumab and other biotherapy entering the market.

The nature of the systemic treatment as well as its administration modalities are defined by the investigator according to usual practice.

All dermatology departments located in the French metropolitan area and using biotherapies as treatment of cutaneous psoriasis will be solicited for participation to the cohort.

The inclusion will last at least 3 years with a follow-up of at least 5 years for each patient (8 years maximum), with a 6 month periodicity for the data collection (complying with good clinical practice for these patients). Follow-up duration may be extended in the case of the identification of safety signals in the early years.

Each study within the cohort has its specific endpoints according to its specific objectives but the whole data required will be collected at the same time for both studies then registered in a single database (eCRF). The statistical analyses will be performed by the clinical investigation and epidemiology center (INSERM CIE 801) of BICHAT hospital's department of epidemiology and clinical research

2 636 patients will be included with the following distribution:.

* Non-exposed group: 1200 patients
* Exposed group: 1436 patients (naive or not) with at least 1200 patients naive for biotherapy.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 years
* Having been informed of the objectives and conduct of the research and having signed a written informed consent to participate
* Consulting or being hospitalized for cutaneous psoriasis (clinical diagnosis) justifying the prescription of a major systemic therapy and for whom cutaneous psoriasis is the main reason for systemic treatment and belonging to one of the two following groups:

  * Patients exposed to a major conventional systemic therapy (methotrexate or cyclosporine, excluding biotherapies) since at least 3 months and for which there are no plans to institute treatment with biotherapy in the next 6 months : non-exposed group.
  * Patients exposed to a biological therapy (infliximab, adalimumab, etanercept, ustekinumab and other biotherapy entering the market) : exposed group.

Exclusion criteria:

* Patients for whom cutaneous psoriasis is not the main reason for systemic treatment: treatment justified by psoriatic arthritis, concomitant Crohn's disease ...;
* Patients unable to comply with the planned cohort monitoring or whose follow-up is expected to be difficult.
* Patient for whom the treatment given at baseline cannot be identified (Patient participating to a double-blind trialinvolving biotherapies for example).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient consulting or being hospitalized for cutaneous psoriasis (clinical diagnosis), justifying the prescription of a major systemic therapy (methotrexate or cyclosporine, or biotherapy) and for whom cutaneous psoriasis is the main reason for systemic treatment
Sampling Method: Non-Probability Sample
Enrollment: 4613 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of skin cancer | Each patient will be followed for at least 5 years(8 years maximum), data being collected at each visit (approximately every 6 month)
  Occurrence of skin cancer (spinocellular carcinomas [including carcinoma in situ (Bowen) and keratoacanthomas], basocellular carcinomas and melanomas).

SECONDARY OUTCOMES:
Event-free survival; incidence of serious adverse events;effectiveness;therapeutic strategy,long-term safety(serious and non-serious adverse events,quality of life, rebounds after treatment discontinuation;maintenance of a therapeutic response over time | Each patient will be followed for at least 5 years(8 years maximum), data being collected at each visit (approximately every 6 month)
  Composite measure

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Chosidow, Md, Phd, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, Île-de-France Region, France